CLINICAL TRIAL: NCT01925755
Title: Prospective Multicenter Observational Non-interventional Local Study on Prescription Behavior of Anticoagulation Therapy in Secondary Stroke Prevention in Atrial Fibrillation Patients
Brief Title: Non-interventional Local Study on Prescription Behavior of Anticoagulation Therapy in Secondary Stroke Prevention in Atrial Fibrillation Patients
Acronym: NEURO-XAR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16627; XA2012-01RU (Other: Company internal)
Record Dates: First submitted 2013-07-15; First posted 2013-08-20 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Stroke; Embolism
Keywords: Non-interventional; Rivaroxaban; Prevention in prior stroke or TIA; Russian Federation
MeSH Terms: conditions — Stroke; Embolism; Ischemic Attack, Transient | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: Rivaroxaban ( Xarelto, BAY59-7939)

INTERVENTIONS:
Other: Rivaroxaban ( Xarelto, BAY59-7939) — Patients with prior stroke or TIA history and who have never taken anticoagulation treatment regarding AF before. One film-coated tablet contains Rivaroxaban 15 mg or 20mg

SUMMARY:
This is local prospective multicenter observational non-interventional local study. Primary study objective is investigate and describe prescription pattern of neurologists in secondary stroke or non-CNS (non-Central Nervous System) systemic embolism prevention in patients with AF (Atrial fibrillation) and prior stroke or TIA (Transient Ischemic attack) who treat with rivaroxaban at an initial visit and three follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years old who start treatment with rivaroxaban
* Non-valvular Atrial Fibrillation is documented in patients' file
* Prior TIA/Stroke history
* TIA - more than 72 hours after documented TIA
* more than 2 weeks after non-hemorrhagic stroke
* Written informed consent

Exclusion Criteria:

* Contraindications for use of Xarelto® in accordance with approved product label
* Previous thromboprophylaxis treatment with anticoagulants prior toby reason of stroke / TIA prevention
* Any reasons of medical and non-medical character, which in the opinion of the physician can hamper patient participation in NIS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients ≥ 18 years old with prior stroke or TIA history and who have never taken anticoagulation treatment regarding AF before and meet criteria of inclusion and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Prescription pattern of neurologists in secondary stroke or non-CNS systemic embolism prevention in patients with AF and prior stroke or TIA who treat with rivaroxaban | up to 6 months
  * Time lag after prior stroke or TIA before Xarelto prescription;
  * Frequency of switching/discontinuation of Xarelto treatment;
  * Time to switching/discontinuation of Xarelto treatment;
  * Reasons of switching/discontinuation of Xarelto treatment (using formalized criteria list);
  * In case of change of treatment - drug, dose, duration of use

SECONDARY OUTCOMES:
Descriptive characteristics of patients after prior stroke/TIA in the need of secondary stroke prevention with Xarelto (gender, age, race, alcohol/smoking, BMI and BP abnormalities, CHA2DS2 VASC, HAS BLED, Rankin Score) | up to 6 months
  CHA2DS2 VASC - Stroke risk assessment scale; HAS BLED - Score for Major Bleeding Risk (in anticoagulation therapy)
Identify time of start of anticoagulation therapy immediately after event (stroke or TIA) for secondary prevention in real life practice | up to 6 months
Describe AE characteristics (frequency, severity, relation to treatment, AE treatment, AE outcome) | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Russia